CLINICAL TRIAL: NCT06687135
Title: The Effectiveness of a Digital Falls Prevention Programme (KOKU) Versus Usual Care to Improve Balance, Falls Risk and Function in Older Adults
Brief Title: Keep-On-Keep-Up (KOKU)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Emma Stanmore, Chief Investigator/ Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PURE ID: 273223769
Record Dates: First submitted 2024-11-04; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-07

CONDITIONS: Balance; Falls Prevention; Functional Decline
Keywords: Balance; Falls Prevention; Functional Decline; Older People; Gerotechnology; Rehabilitation

STUDY DESIGN:
Intervention Model Description: A two-arm randomised controlled trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KOKU (Experimental): A maximum of 196 participants will be recruited to participate in the study, across sites in Greater Manchester and Lancashire, UK.
  Participants will be randomised into either;
  * the experimental group (n=98); who will receive the KOKU intervention or
  * the control group (n=98); who will receive the FaME/ OTAGO exercise and falls prevention information leaflets without KOKU.
  Interventions: Other: KOKU
- FaME/OTAGO (Active Comparator): A maximum of 196 participants will be recruited to participate in the study, across sites in Greater Manchester and Lancashire, UK.
  Participants will be randomised into either;
  * the experimental group (n=98); who will receive the KOKU intervention or
  * the control group (n=98); who will receive the FaME/ OTAGO exercise and falls prevention information leaflets without KOKU.
  Interventions: Other: FaME / OTAGO leaflet and AGE UK Stay Steady Leaflet

INTERVENTIONS:
Other: KOKU — KOKU is a digital strength and balance programme designed to prevent physical decline and frailty KOKU provides access to personalised, progressive strength and balance exercises.
  More information can be found at: https://kokuhealth.com/
  Other Names: Keep-On-Keep-Up
  Arms: KOKU
Other: FaME / OTAGO leaflet and AGE UK Stay Steady Leaflet — A leaflet with information on a combination of strength and balance exercises and walking programs, performed on a weekly basis by older adults at home, or community settings. The exercises can be done individually or in a group setting and are aimed at reducing falls in older adults.
  More information can be found at: https://fameexercise.com/ and https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf https://www.ageuk.org.uk/information-advice/health-wellbeing/exercise/staying-steady-download-page/#:~:text=This%20guide%20outlines%20things%20you%20can
  Other Names: Fitness-and-Mobility-Exercises (FaME) / OTAGO-Exercise-Program (OEP) and AGE UK Stay Steady Leafletleaflets
  Arms: FaME/OTAGO

SUMMARY:
Falls are the primary cause of fatal and non-fatal accidental injuries in older adults. Around a third of community-dwelling older adults fall per year with high associated personal and societal costs. The World Falls Prevention Guidelines recommend balance challenging, functional exercise programmes for falls prevention but there can be low uptake and adherence in community settings. A digital, NHS approved programme Keep-On-Keep-Up (KOKU) was co-developed with older adults and therapists, to provide progressive, evidence-based exercises and to raise awareness of home hazards and ways to improve bone health, nutrition and hydration. This trial aims to investigate the effectiveness of the KOKU digital strength and balance programme for improving balance, function and reducing falls risk in community dwelling older adults.

Objective:

The purpose of this study is to investigate the effectiveness and cost-effectiveness of an NHS (National Health Service) approved, digital falls prevention intervention; (Keep On Keep Up (KOKU) - see https://kokuhealth.com) for improving balance, maintaining function and reducing falls risk in community dwelling older adults.

Design:

A two-arm randomised controlled trial.

Participants and setting:

Community-dwelling older adults aged 65 years and older.

Interventions:

Digital 12-week strength and balance programme, plus standard care (falls prevention exercises advice and leaflet) against standard care only.

Main outcome measures:

The primary outcome measure is balance function at 12 weeks post-baseline, as assessed by the Berg Balance scale (BBS). Secondary outcomes include: healthcare utilisation and health-related quality of life, fear of falling, mobility, self-reported physical activity, falls risk, pain, mood, fatigue, and self-reported falls over a 3-month period. Randomisation will take place after participants are recruited and baseline data is collected.

DETAILED DESCRIPTION:
* Eligible participants will be advised to use KOKU (a digital health wellbeing app) three times per week for 20-30 minutes
* The KOKU intervention will run for 12 weeks to test the effectiveness
* The control group will be given FaME/ OTAGO exercise and falls prevention information leaflets without KOKU
* Assessments will take place at baseline, 6 weeks, and at the end of the12-week period
* Outcome measures to be used include a series of standardised tests and questionnaires and each participant will be aided in completing these measures
* At the end of the 12 weeks, focus groups and interviews will be conducted to assess the care managers, carers and participant's perspectives regarding the effectiveness of the KOKU digital program and its usability

ELIGIBILITY:
Inclusion Criteria:

* Older adults (aged 60 years and older, inclusive of all genders and ethnicities)
* Are able and willing to provide informed consent (to participate in the study)
* Are able to understand and speak English (to communicate with researchers and understand what the research involves)
* Are able to see and safely use the tablet-based program and read instructions with or without glasses as assessed by the trained research staff (in order to access the intervention)

Exclusion Criteria:

* Inability to understand the study procedures
* Currently using other digital technologies to exercise (would not be a true experimental or control group participant)
* Medical contraindications to exercise e.g. acute illness, severe congestive cardiac failure, uncontrolled hypertension, recent fracture or surgery; myocardial infarction or stroke in past 6 months; severe cognitive impairment; orthopaedic surgery in last 6 months, or on waiting list to have orthopaedic surgery; wheelchair users; severe auditory or visual impairment; and peripheral neuropathy or other uncontrolled medical (conditions that are likely to compromise the ability to exercise)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  The primary outcome measure is balance function as measured by the Berg Balance Scale (BBS). The BBS is a 14-item scale designed to measure balance of the older adult in a clinical setting. Each item consists of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. The total score equals 56. Score of < 45 indicates individuals may be at greater risk of falling (Berg et al., 1992).

SECONDARY OUTCOMES:
European Quality of Life 5 Dimensions (EQ5D-5L) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  The 5-level EQ-5D version (EQ-5D-5L) measures health-related quality of life and consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient selects the most appropriate statement in each of the five dimensions which results in a 1-digit number for the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Higher scores indicate better health-related quality of life. Minimum score is -0.285 and maximum score is 1.
5-item Geriatric Depression Scale (GDS) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  Mood will be assessed using the 5-item Geriatric Depression Scale (GDS). This screening tool for depression in older adults is validated for older adults in a wide range of settings (Hoyl et al., 1999). The scale ranges from minimum score of 0 indicating no depression to 5 indicating higher level of depressive symptoms.
Physical Activity Scale for the Elderly (PASE) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess the participant's physical activity levels. The PASE score theoretically ranges from 0 indicating no physical activity to a maximum score of over 400 (depending on the intensity, frequency and duration of the activities) indicating greater levels of physical activity.
Short Falls Efficacy Scale-International (FES-I) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess confidence in performing activities of daily living without falling.(concerns about falling). The scale ranges from 7 to 28 with 7 as the minimum score indicating no concerns about falling and 28 is the maximum score indicating severe concern about falling.
Five times Sit to Stand Test | Baseline, 6 weeks and 12 weeks
  The 5-times Sit-to-Stand Test assesses lower body strength, lower limb power, and functional mobility. It measures the time in seconds taken to complete five consecutive sit-to-stand movements as quickly as possible from a seated position. There are no fixed minimum or maximum scores in time, higher scores indicate worse performance. For older adults a time greater than 12 seconds is often used as a threshold indicating an increased risk of falls or mobility limitations.
Assessment of Falls Risk Tool (FRAT) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess risk of falls, 0 is the minimum score indicating no or very low risk of falls and 20 is the maximum score indicating a very high risk of falls.
System Usability Scale (SUS) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess the usability of KOKU. The SUS provides a score between 0 and 100 with 0 the minimum score indicating poor usability and 100 the maximum score indicating excellent usability.
Theoretical Framework for Acceptability (TFA) | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess the usability of KOKU. The TFA is reported qualitatively to capture a detailed understanding of acceptability in healthcare settings.
12 Item Short Scale for Measuring Technology Commitment | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess the usability of KOKU. The 12 Item Short Scale for Measuring Technology Commitment follows a likert-type scale (ranging 1 to 5 for each item). The total score is then calculated by summing the items. The minimum score is 12 representing the lowest commitment to technology and the maximum score is 60 indicating highest level of commitment to technology.
The Short Version of the User Experience Question | 0 Weeks (baseline), 6 weeks and 12 weeks (study completion)
  To assess the usability of KOKU. The Short Version of the User Experience Question (UEQ) is composed of 6 dimensions of user experience (attractiveness, efficiency, perspicuity, dependability, stimulation and novelty) rated on a 7 point Likert scale ranging from 1 to 7. The minimum score is 6 indicating low user experience and the maximum score is 42 indicating high user experience.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Stanmore, PhD, Principal Investigator — The University of Manchester
Locations (2):
- United Kingdom (2):
  - The University of Manchester, Manchester, Greater Manchester
  - University of Manchester, Manchester, Greater Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Keep On Keep Up (KOKU) — https://kokuhealth.com/
- See also: Fitness and Mobility Exercises (FaME) — https://fameexercise.com/
- See also: OTAGO Exercise Programme (OEP) — https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf